CLINICAL TRIAL: NCT01156961
Title: Post Registration Observational Program for Patients With Locally Recurrent or Metastatic Breast Cancer Who Receive Bevacizumab (Avastin) in Combination With Paclitaxel for the First-line Treatment
Brief Title: A Study of The Safety Profile of First-line Avastin (Bevacizumab) in Combination With Paclitaxel in Patients With Locally Recurrent or Metastatic Her2-negative Breast Cancer (AVATAX)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Absence of patient's recruitment in the study due to administrative reasons
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25081
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: paclitaxel

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 10 mg/kg iv every 2 weeks or 15 mg/kg iv every 3 weeks
Drug: paclitaxel — 90 mg/m2 iv days 1, 8 and 15 of every 28-day cycle or 175 mg/m2 iv day 1 of each 21-day cycle

SUMMARY:
This single arm, open label study will assess the safety profile of Avastin (bevacizumab) in combination with paclitaxel as first-line treatment in patients with locally recurrent or metastatic Her2-negative breast cancer. Patients will receive Avastin, either 10 mg/kg intravenously (iv) every 2 weeks or 15 mg/kg iv every 3 weeks. Correspondingly, paclitaxel will be administered at a dose of 90 mg/m2 o days 1, 8 and 15 of every 28-day cycle or 175 mg/m2 on day 1 of every 21-day cycle. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Locally recurrent or metastatic Her2-negative breast cancer
* Locally recurrent disease must not be amenable to radiation therapy or resection with curative intent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Prior Adjuvant chemotherapy allowed; if taxane-based a disease-free interval after completion of >/=12 months is required
* Adequate haematological, renal and liver function

Exclusion Criteria:

* Previous chemotherapy for locally recurrent or metastatic disease
* Radiation therapy for metastatic disease (except for relief of metastatic bone pain with irradiation of </= 30% of marrow-bearing bone)
* CNS metastases
* Pre-existing peripheral neuropathy
* Clinically significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Safety profile: Adverse events | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche